CLINICAL TRIAL: NCT02562755
Title: A Phase 3 Randomized, Open-Label Study Comparing Pexa Vec (Vaccinia GM CSF / Thymidine Kinase-Deactivated Virus) Followed by Sorafenib Versus Sorafenib in Patients With Advanced Hepatocellular Carcinoma (HCC) Without Prior Systemic Therapy
Brief Title: Hepatocellular Carcinoma Study Comparing Vaccinia Virus Based Immunotherapy Plus Sorafenib vs Sorafenib Alone
Acronym: PHOCUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SillaJen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JX594-HEP024
Record Dates: First submitted 2015-09-24; First posted 2015-09-29 (Estimated); Results first posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Hepatocellular Carcinoma (HCC); Pexastimogene Devacirepvec (Pexa-Vec); Sorafenib; GM-CSF therapy; Thymidine Kinase-Deactivated Vaccinia Virus; Oncology; Recombinant Vaccinia Virus; Oncolytic Virus Therapy; Oncolytic virotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasms; Vaccinia | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pexa-Vec followed by Sorafenib (Experimental): Pexa-Vec (pexastimogene devacirepvec) will be administered as 3 bi-weekly intratumoral (IT) injections of 1e9 pfu at day 1 and weeks 2 and 4, followed by sorafenib at Week 6.
  Interventions: Biological: Pexastimogene Devacirepvec (Pexa Vec); Drug: Sorafenib
- Sorafenib (Active Comparator): Sorafenib (400 mg twice daily) begins on Day 1.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Biological: Pexastimogene Devacirepvec (Pexa Vec) — Pexa-Vec is a vaccinia virus based oncolytic immunotherapy designed to stimulate the immune system following infection and replication within tumor cells.
  Other Names: JX-594
  Arms: Pexa-Vec followed by Sorafenib
Drug: Sorafenib — Sorafenib belongs to the pharmacotherapeutic group of antineoplastic agents, protein kinase inhibitors, ATC code: L01XE05.
  Sorafenib is a multi-kinase inhibitor which has demonstrated both anti-proliferative and anti-angiogenic properties in vitro and in vivo.
  Sorafenib is approved for the treatment of advanced HCC and is the Standard Of Care for this disease.
  Other Names: Nexavar

SUMMARY:
This is a randomized Phase 3 study to determine whether treatment with vaccinia virus based immunotherapy (Pexa-Vec) followed by sorafenib increases survival compared to treatment with sorafenib in patients with advanced hepatocellular carcinoma who have not received prior systemic therapy.

DETAILED DESCRIPTION:
This is a multi-center, randomized, open-label, Phase 3 study comparing Pexa Vec followed by sorafenib versus sorafenib in patients with advanced HCC without prior systemic therapy.

A total of 459 patients were randomly assigned to 2 treatment arms- 234 patients in the Pexa-Vec followed by sorafenib treatment group and 225 patients in the sorafenib only treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Histological/cytological diagnosis of primary HCC
* Advanced stage HCC (Barcelona Clinic Liver Cancer [BCLC] Stage C or B per American Association for the Study of Liver Disease [AASLD] guidelines)
* At least one measurable viable tumor in the liver, ≥1 cm longest diameter (LD), using a dynamic imaging technique (arterial phase of triphasic computerized tomography [CT] scan, or dynamic contrast-enhanced magnetic resonance imaging [MRI]), and injectable under imaging-guidance (CT and/or ultrasound)
* Child-Pugh Class A
* Performance status 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale
* Adequate hematological, hepatic, and renal function:
* Additional inclusion criteria exist

Exclusion Criteria:

* Histological diagnosis of cholangiocarcinoma, hepatocholangiocarcinoma, fibrolamellar carcinoma and hepatoblastoma
* Symptomatic cardiovascular disease, including but not limited to significant coronary artery disease (e.g., requiring angioplasty or stenting) or congestive heart failure within the preceding 12 months
* Current or past history of cardiovascular disease (e.g.. past history of myocardial infarction, ischemic cardiomyopathy) unless cardiology consultation and clearance has been obtained for study participation
* History of moderate or severe ascites, bleeding esophageal varices, hepatic encephalopathy or pleural effusions related to liver insufficiency within 6 months of screening
* Bulky disease patients - tumors encompassing >50% of the liver volume and / or inferior vena cava invasion
* Known significant immunodeficiency due to underlying illness (e.g., HIV/AIDS) and/or immune-suppressive medication including high-dose corticosteroids
* Ongoing severe inflammatory skin condition (as determined by the Investigator) requiring medical treatment
* History of severe eczema (as determined by the Investigator) requiring medical treatment
* Additional exclusion criteria exist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SillaJen Medical, Study Director — SillaJen, Inc.
Locations (142):
- United States (23):
  - University of Alabama, Birmingham, Alabama
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - UC Irvine Medical Center, Orange, California
  - Stanford University School of Medicine, Palo Alto, California
  - University of Florida Shands Hospital, Gainesville, Florida
  - University of Chicago, Chicago, Illinois
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Mercy Medical Center, Inc., Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Kansas City Research Institute, Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - Morristown Medical Center, Morristown, New Jersey
  - St. Joseph's Hospital, Paterson, New Jersey
  - Ohio State University, Columbus, Ohio
  - Hospital of The University of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Benaroya Research Institute at Virginia Mason Hospital, Seattle, Washington
- Australia (13):
  - Site No. 8409, Adelaide
  - Site No. 8412, Adelaide
  - Site No. 8403, Brisbane
  - Site No. 8401, Camperdown
  - Site No. 8407, Clayton
  - Site No. 8406, Concord
  - Site No. 8408, Fitzroy
  - Site No. 8405, Footscray
  - Site No. 8414, Heidelberg
  - Site No. 8411, Melbourne
  - Site No. 8402, Parkville
  - Site No. 8415, Perth
  - Site No. 8413, Sydney
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
- China (19):
  - Site 8829, Changchun
  - Site No. 8821, Changsha
  - Site 8811, Fuzhou
  - Site 8820, Fuzhou
  - Site No.8816, Guangdong
  - Site 8827, Guangzhou
  - Site No.8828, Guangzhou
  - Site 8832, Hangzhou
  - Site No. 8802, Harbin
  - Site 8805, Hefei
  - Site No. 8808, Hefei
  - Site No.8815, Hefei
  - Site No. 8801, Nanjing
  - Site 8833, Qingdao
  - Site 8806, Shanghai
  - Site 8822, Shanghai
  - Site 8831, Shanghai
  - Site No. 8823, Xi'an
  - Site No. 8825, Xi'an
- France (13):
  - Site No. 9013, Bondy
  - Site No. 9005, Bordeaux
  - Site No. 9003, Créteil
  - Site No. 9006, Lille
  - Site 9012, Montpellier
  - Site No. 9008, Nantes
  - Site No. 9010, Nice
  - Site No. 9007, Paris
  - Site No. 9014, Paris
  - Site No. 9011, Rennes
  - Site No. 9001, Strasbourg
  - Site No. 9002, Toulouse
  - Site No. 9009, Vandœuvre-lès-Nancy
- Germany (11):
  - Site No. 9111, Aachen
  - Site No. 9113, Bonn
  - Site No. 9109, Dresden
  - Site No. 9108, Frankfurt am Main
  - Site No. 9106, Hamburg
  - Site No 9105, Hannover
  - Site No. 9112, Heidelberg
  - Site No. 9101, Mainz
  - Site No. 9102, München
  - Site No. 9104, Tübingen
  - Site No. 9110, Ulm
- Site No. 8601, Hong Kong, Hong Kong
- Israel (6):
  - Site No. 9707, Afula
  - Site 9704, Haifa
  - Site No. 9702, Haifa
  - Site No. 9705, Jerusalem
  - Site No. 9703, Ramat Gan
  - Site No. 9706, Tel Aviv
- Italy (4):
  - Site No.9205, Modena
  - Site No. 9204, Napoli
  - Site No. 9201, Palermo
  - Site No. 9203, Parma
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Site No. 8902, Christchurch
- Portugal (5):
  - Site No. 9404, Coimbra
  - Site No. 9405, Coimbra
  - Site No. 9403, Lisbon
  - Site No. 9401, Porto
  - Site No. 9402, Porto
- Singapore (3):
  - Site 8702, Singapore
  - Site 8703, Singapore
  - Site No. 8701, Singapore
- South Korea (21):
  - Site No. 8208, Ansan
  - Site No. 8211, Bucheon-si
  - Site No. 8201, Busan
  - Site 8216, Daegu
  - Site No. 8207, Daegu
  - Site No. 8213, Daegu
  - Site No. 8220, Daegu
  - Site 8224, Goyang
  - Site No. 8221, Jinju
  - Site No. 8218, Pusan
  - Site No. 8222, Seongnam
  - Site No. 8219, Seongnam-si
  - Site No. 8202, Seoul
  - Site No. 8203, Seoul
  - Site No. 8205, Seoul
  - Site No. 8209, Seoul
  - Site No. 8212, Seoul
  - Site No. 8215, Seoul
  - Site No. 8223, Seoul
  - Site No. 8210, Suwon
  - Site No. 8217, Ulsan
- Taiwan (6):
  - Site No. 8305, Kaohsiung City
  - Site No. 8307, Linkou District
  - Site No. 8306, Taichung
  - Site No. 8302, Tainan
  - Site No. 8301, Taipei
  - Site No. 8303, Taipei
- Thailand (6):
  - Site No. 8502, Bangkok
  - Site No. 8505, Bangkok
  - Site No. 8503, Chiang Mai
  - Site No. 8507, Hat Yai
  - Site No. 8501, Khon Kaen
  - Site No. 8506, Phitsanulok
- United Kingdom (6):
  - Site No. 9501, Birmingham
  - Site No. 9505, Guildford
  - Site No. 9503, Leeds
  - Site No. 9502, London
  - Site No. 9504, London
  - Site No. 9506, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pexa-Vec Followed by Sorafenib: Pexa-Vec (pexastimogene devacirepvec) will be administered as 3 bi-weekly intratumoral (IT) injections of 1e9 pfu at day 1 and weeks 2 and 4, followed by sorafenib at Week 6.
  Pexastimogene Devacirepvec (Pexa Vec): Pexa-Vec is a vaccinia virus based oncolytic immunotherapy designed to stimulate the immune system following infection and replication within tumor cells.
  Sorafenib: Sorafenib belongs to the pharmacotherapeutic group of antineoplastic agents, protein kinase inhibitors, ATC code: L01XE05.
  Sorafenib is a multi-kinase inhibitor which has demonstrated both anti-proliferative and anti-angiogenic properties in vitro and in vivo.
  Sorafenib is approved for the treatment of advanced HCC and is the Standard Of Care for this disease.
- Sorafenib: Sorafenib (400 mg twice daily) begins on Day 1.
  Sorafenib: Sorafenib belongs to the pharmacotherapeutic group of antineoplastic agents, protein kinase inhibitors, ATC code: L01XE05.
  Sorafenib is a multi-kinase inhibitor which has demonstrated both anti-proliferative and anti-angiogenic properties in vitro and in vivo.
  Sorafenib is approved for the treatment of advanced HCC and is the Standard Of Care for this disease.
Period: Overall Study
Arm/Group | Pexa-Vec Followed by Sorafenib | Sorafenib
Started (Randomized) | 234 | 225
Safety Population (Patients who received at least one dose of study treatment) | 218 | 217
Completed | 161 | 153
Not Completed | 73 | 72

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pexa-Vec Followed by Sorafenib | Sorafenib | Total
Number analyzed (Participants) | 234 | 225 | 459
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 133 | 148 | 281
  >=65 years | 101 | 77 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (10.05) | 60.5 (11.06) | 60.9 (10.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 43 | 73
  Male | 204 | 182 | 386
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 229 | 219 | 448
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Singapore | 8 | 3 | 11
  Hong Kong | 1 | 3 | 4
  United States | 40 | 34 | 74
  United Kingdom | 3 | 4 | 7
  Thailand | 2 | 5 | 7
  Portugal | 2 | 3 | 5
  New Zealand | 27 | 27 | 54
  Canada | 5 | 4 | 9
  South Korea | 61 | 68 | 129
  China | 42 | 40 | 82
  Taiwan | 13 | 10 | 23
  Italy | 1 | 3 | 4
  Israel | 1 | 2 | 3
  Australia | 9 | 5 | 14
  France | 12 | 8 | 20
  Germany | 7 | 6 | 13
ECOG performance status [Count of Participants; unit: Participants] — The ECOG Performance Status describes a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.): Grade 0, Fully active, able to carry on all pre-disease performance without restriction; Grade 1, Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  Participants
    0 | 146 | 142 | 288
    1 | 88 | 83 | 171

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Percentage of participants who showed overall response during their participation in the study. Per Modified Response Evaluation Criteria In Solid Tumors Criteria (mRECIST) and assessed by tri-phasic contrast enhanced CT: Complete Response (CR), Disappearance of intratumoral enhancing area; Partial Response (PR), >=30% decrease in the sum of the diameters of enhancing area; Overall Response (OR) = CR + PR.
Time Frame: From date of randomization to the date of first documented radiographic tumor progression up to 53 months
Measure: Number; unit: percentage of participants
Arm/Group | Pexa-Vec Followed by Sorafenib | Sorafenib
Number analyzed (Participants) | 234 | 225
percentage of participants | 19.2 | 20.9

ADVERSE EVENTS:
Time Frame: From date of randomization to end of participation in the study, up to 53 months
Arm/Group | Pexa-Vec Followed by Sorafenib | Sorafenib
All-Cause Mortality (participants affected / at risk) | 33/218 | 25/217
Serious Adverse Events (participants affected / at risk) | 117/218 | 77/217
Other Adverse Events (participants affected / at risk) | 218/218 | 214/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pexa-Vec Followed by Sorafenib (N=218) | Sorafenib (N=217)
Hypotension (Vascular disorders) | 2 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Liver carcinoma ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anaphylactic Reaction (Immune system disorders) | 0 | 1
Pyrexia (General disorders) | 8 | 1
Asthenia (General disorders) | 3 | 5
General physical health deterioration (General disorders) | 2 | 1
Fatigue (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 2 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Death NOS (General disorders) | 1 | 0 — Death Not Otherwise Specified
Confusional state (Psychiatric disorders) | 1 | 0
Hepatic rupture (Injury, poisoning and procedural complications) | 3 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Blood bilirubin increased (Injury, poisoning and procedural complications) | 1 | 4
Aspartate aminotransferase increased (Injury, poisoning and procedural complications) | 2 | 0
Blood creatinine increased (Injury, poisoning and procedural complications) | 0 | 1
Angina pectoris (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0
Aortic valve disease (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Atrial thrombosis (Cardiac disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 4 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 5 | 4
Ischaemic stroke (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Alcoholic seizure (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 7 | 3
Ascites (Gastrointestinal disorders) | 8 | 4
Abdominal pain (Gastrointestinal disorders) | 4 | 5
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 1
Constipation (Gastrointestinal disorders) | 2 | 2
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 1
Haematemesis (Gastrointestinal disorders) | 2 | 0
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 1
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 4 | 3
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 11 | 8
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 3 | 0
Bile duct stenosis (Hepatobiliary disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 2 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 1
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Biliary dilatation (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 2 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatic haemorrhage (Hepatobiliary disorders) | 2 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 1
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Gout (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 4
Sepsis (Infections and infestations) | 1 | 4
Peritonitis bacterial (Infections and infestations) | 4 | 0
Liver abscess (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Pneumonia necrotising (Infections and infestations) | 1 | 0
Mycobacterial infection (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Rectal abscess (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Hepatitis viral (Infections and infestations) | 0 | 1
Dengue fever (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Paraplegia (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pexa-Vec Followed by Sorafenib (N=218) | Sorafenib (N=217)
Hypertension (Vascular disorders) | 44 | 39
Hypotension (Vascular disorders) | 35 | 2
Pyrexia (General disorders) | 184 | 28
Fatigue (General disorders) | 65 | 64
Chills (General disorders) | 71 | 4
Asthenia (General disorders) | 22 | 21
Influenza like illness (General disorders) | 37 | 5
Injection site pain (General disorders) | 27 | 0
Insomnia (Psychiatric disorders) | 16 | 20
Procedural pain (Injury, poisoning and procedural complications) | 12 | 2
Weight decreased (Investigations) | 58 | 49
Aspartate aminotransferase increased (Investigations) | 30 | 39
Blood bilirubin increased (Investigations) | 22 | 33
Alanine aminotransferase increased (Investigations) | 17 | 29
Platelet count decreased (Investigations) | 15 | 15
Sinus tachycardia (Cardiac disorders) | 13 | 3
Tachycardia (Cardiac disorders) | 16 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 31 | 25
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 | 10
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 10 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 | 9
Anaemia (Blood and lymphatic system disorders) | 33 | 23
Headache (Nervous system disorders) | 33 | 23
Dizziness (Nervous system disorders) | 20 | 13
Diarrhoea (Gastrointestinal disorders) | 107 | 116
Nausea (Gastrointestinal disorders) | 74 | 63
Abdominal pain (Gastrointestinal disorders) | 62 | 60
Constipation (Gastrointestinal disorders) | 52 | 51
Vomiting (Gastrointestinal disorders) | 56 | 27
Ascites (Gastrointestinal disorders) | 46 | 36
Abdominal pain upper (Gastrointestinal disorders) | 43 | 30
Abdominal distension (Gastrointestinal disorders) | 26 | 26
Stomatitis (Gastrointestinal disorders) | 17 | 24
Dyspepsia (Gastrointestinal disorders) | 15 | 13
Palmar plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 73 | 99
Alopecia (Skin and subcutaneous tissue disorders) | 32 | 46
Rash (Skin and subcutaneous tissue disorders) | 23 | 28
Pruritus (Skin and subcutaneous tissue disorders) | 16 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 | 12
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14 | 12
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 8
Decreased appetite (Metabolism and nutrition disorders) | 85 | 64
Hypokalaemia (Metabolism and nutrition disorders) | 18 | 19
Hypoalbuminaemia (Metabolism and nutrition disorders) | 15 | 11
Hyponatraemia (Metabolism and nutrition disorders) | 16 | 10
Hyperkalaemia (Metabolism and nutrition disorders) | 14 | 4
Rash pustular (Infections and infestations) | 39 | 2
Upper respiratory tract infection (Infections and infestations) | 17 | 23
edema peripheral (General disorders) | 27 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/55/NCT02562755/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT02562755/SAP_001.pdf